CLINICAL TRIAL: NCT02511756
Title: Visualization of Anti-angiogenic Effects With Perfusion Computed Tomography (CTP) in mCRC Patients Treated With First-line Bevacizumab
Brief Title: Visualization of Anti-angiogenic Effects With Perfusion Computed Tomography (CTP)
Acronym: AVA-CTP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Patrick Veit-Haibach (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Patrick Veit-Haibach, PD MD, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2015-0084
Record Dates: First submitted 2015-04-29; First posted 2015-07-30 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Perfusion-computed tomography
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tomography Scanners, X-Ray Computed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perfusion-computed tomography (CTP) (Other): Patients undergo a total of four perfusion-computed tomographies from baseline to progression of disease.
  Interventions: Device: Computed tomography X-ray system

INTERVENTIONS:
Device: Computed tomography X-ray system — Contrast-enhanced computed tomography of liver metastases
  Other Names: CT scanner

SUMMARY:
The primary objective of this study is to investigate the anti-angiogenic effect of bevacizumab measured by CTP as a predictive marker for efficacy measured by progression-free survival (PFS) in mCRC patients under first-line bevacizumab-containing, fluoropyrimidine-based chemotherapy

DETAILED DESCRIPTION:
So far, CTP has provided non-invasive imaging of tumor biological response to anti-angiogenic and vascular targeting agents in a number of clinical trials with increasing clinical application. CTP can be examined with a variety of commercially available CE-certified CT scanners and imaging post-processing is possible with commercially available CE-certified software from different vendors, too. In several studies, anti-angiogenic effects have been detected with CTP but further evidence for its clinical validation has to be proven in clinical trials.

Changes in tumor vasculature measured by CTP will be correlated to the clinical efficacy parameters progression-free survival, overall survival and response rate, thus identifying a group of patients who profit most from the anti-angiogenic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, male or female
* Signed written informed consent
* Patients with histologically confirmed diagnosis of colorectal cancer with hepatic metastases who are candidates for systemic treatment.
* Confirmation of metastatic liver disease within one month prior to inclusion in one of the following radiological procedures:

  * Contrast-enhanced spiral computed tomography showing at least one liver nodule ≥ 20 mm in longest diameter according to RECIST 1.1 criteria
  * MR imaging of the liver with liver lesions suspicious for metastases
  * PET computed tomography (PET/CT) with liver lesions suspicious for metastases
* Patient is eligible and designated for treatment with standard-of-care first-line bevacizumab-containing, fluoropyrimidine-based chemotherapy.
* ECOG performance status ≤ 2 (see appendix)

Exclusion Criteria:

* Inability or unwillingness to comply with the participation requirements
* History of untreated hyperthyreosis
* History of intolerance of or allergy to iodine contrast media according to CTCAE V4.03
* Calculated creatinine clearance < 45 ml/min
* For fertile women: positive urine pregnancy test or lactation.
* Known or suspected non-compliance, drug or alcohol abuse
* Life expectancy of less than 3 months
* Participation in another interventional trial with an investigational medicinal product (IMP) and within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
CTP as predictive marker for efficacy measured by progression-free survival | one year
  Predictive power of decrease in tumor vasculature on the clinical outcome in bevacizumab-based chemotherapy measured by progression-free survival (PFS). Decrease in tumor vasculature is measured by blood flow in CTP 3 compared to CTP 1 (baseline)

SECONDARY OUTCOMES:
CTP as predictive marker for efficacy measured by progression-free survival | one year
  Predictive power of decrease in tumor vasculature on the clinical outcome in bevacizumab-based chemotherapy measured by progression-free survival (PFS). Decrease in tumor vasculature is measured by blood flow, blood volume, mean transit time and permeability surface-area product in CTP
CTP as predictive marker for efficacy measured by overall survival | four years
  Predictive power of decrease in tumor vasculature measured by CTP on the clinical outcome in bevacizumab-based chemotherapy measured by overall survival (OS)
Tumor vasculature at progression | one year
  Tumor vasculature measured by blood flow, blood volume, mean transit time and permeability surface-area product in CTP at the time of confirmed progression
Subgroup analyses according to the RAS mutation status, BRAF mutation status and VEGF-A level | one year
  Predictive power of RAS-mutation status, BRAF-mutation status and VEGF-A level on the clinical outcome in bevacizumab-based chemotherapy measured by progression-free survival (PFS)
Local and distant recurrences | one year
  Rates of local and distant recurrences according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Hospital Zurich, Diagnostic and Interventional Radiology
Locations (5):
- Switzerland (5):
  - Luzerner Kantonsspital, Lucerne, Canton of Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Universitätsspital Zürich, Zurich, Canton of Zurich
  - Kantonsspital Graubünden, Chur, Kanton Graubünden